# Inter-rater Reliability of the Clinical Frailty Scale in a Swedish Emergency Department setting

03/30/2021

### **Subject study information**

We would like to ask you to participate in a research project. In this document, you will be informed about the project and what it means to participate

#### What kind of project is this, and why do you want me to participate?

Clinical Frailty Scale (CFS) is an instrument that assesses the degree of frailty of an older person. CFS can be used in clinical work in an emergency department (ED) and has been evaluated to some extent regarding the degree of observer agreement when the same assessors assess the same patient (inter-rater reliability). However, it has never been studied in a Swedish ED, which is why the purpose of this study is to evaluate the inter-rater reliability of CFS when it is used in clinical work in Swedish ED:s.

At the same time, Loss of Independence (LoI = inability to rise with or without help) has proven to be a possible, simple and cost effective tool to predict risk of mortality and hospitalisation.

For LoI, there is still no information on how high the agreement between different assessors is, which is why we now want to investigate it in this study.

You are asked now to participate in these studies, as you are part of the care team who are responsible for a patient to be assessed regarding degree of frailty and inability to rise with or without assistance.

#### How will this study be done?

You will make an individual assessment of the patient's frailty using the CFS and LoI, as do other team members. You make the assessment just as usual and have access to the usual patient data. What differs from routine is that **you and the other team members perform one assessment each**, and **should not have knowledge of each other's assessments**. The time for each assessment will also be measured with a timer to collect data regarding how time consuming the various assessment-tool are.

#### What happens with the information about me?

The project will collect and register information about you. The information collected is what you state on the work sheet, i.e. your points for the patient's frailty, your HSA-ID, your professional role, number of working years and your age and gender. The information will not be able to be traced to you in the result. Your answers and results will be processed so that unauthorised persons cannot take part in them.

Information that can be linked to you in this way is counted as personal data in accordance with the EU Data Protection Regulation 2016/679 (GDPR). The reason why the project needs to process such personal data is to be able to describe the group that was studied in the research project, your HSA ID is needed to identify your answers in case you wish to cancel your participation in the study.

Region Östergötland is responsible for processing the data. According to the EU Data Protection Regulation, Article 6.1, the legal basis for the processing of personal data is the general interest of research.

Only authorised researchers in the project will be given access to the personal data. When the project is completed, what has been collected and processed within the project will be stored for at least ten years in the Emergency departments local archive or at the regional archive in Region Östergötland.

According to the EU Data Protection Regulation, you have the right to access the information about you that is handled in the study free of charge, and if necessary get any errors corrected. You can also request that information about you be deleted and that the processing of your personal data be restricted. However, the right to delete and restrict the processing of personal data does not apply when the data is necessary for the research in question. If you want to take part in the information, you must contact the principal researcher. The Data Protection Officer can be reached at dataskyddsombud@regionostergotland.se. If you are dissatisfied with how your personal data is processed, you have the right to lodge a complaint with the Privacy Protection Authority, which is the supervisory authority.

#### How do I get information about the results of the study?

The results from the study will be published in a scientific journal, but also internally at the emergency department as the study evaluates instruments that according to the decision will be implemented in quality improvement work. The results will be presented at group level, without the possibility of tracking any individual.

#### **Participation is voluntary**

Your participation is voluntary and you can choose to cancel your participation at any time. If you choose not to participate or want to cancel your participation, you do not have to state why, nor will it affect you at your workplace. If you wish to cancel your participation, please contact the person responsible for the study (see below).

#### Responsibility for the study

Responsible for the study is Region Östergötland, 581 91 Linköping, 010-103 00 00, Principal Investigator is Docent Daniel Wilhelms, Akutkliniken US, daniel.wilhelms@liu.se Contact

Evaluation of an instrument for frailty assessment in Swedish emergency departments

person is Clinical Nurse Specialist Erika Hörlin, Akutkliniken US, erika.horlin@regionostergotland.se

Evaluation of an instrument for frailty assessment in Swedish emergency departments

## Consent to participate in the study

| I have received oral and written information regarding the study and has had the opportunity to ask questions. I may keep the written information. | | |
|---|---|---|
| | ☐ I consent to participate in the study Evaluation of an instrument for frailty assessment in Swedish emergency departments. | |
| ☐ I agree that information about me is processed in the manner described in the research person's information. | | |
| Location and date | | Participants signature |